CLINICAL TRIAL: NCT02584920
Title: A Pharmacokinetic and Pharmacodynamic Study Comparing HLX01 And Rituximab in Patients With CD20-Positive, B-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX01-NHL02
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: B-cell Non Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HLX01 (Experimental): 375mg/m2 iv single dose
  Interventions: Drug: HLX01
- Rituximab (Active Comparator): 375mg/m2 iv single dose
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: HLX01
  Arms: HLX01
Drug: Rituximab
  Arms: Rituximab

SUMMARY:
Randomised, double-blind, parallel group study to compare PK and PD profiles between HLX01 and rituximab (MabThera®) in patients with CD20+ B-cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. aged from 18 to 65 years;
2. CD20-positive non-Hodgkin's lymphoma (NHL);
3. having obtained CR (complete remission) or CRu (uncertain complete remisson) after the prior therapy;
4. ECOG performance status of <=1, expected survival of at least >= 3 months;
5. Peripheral blood lymphocyte count < 5×10^9/L
6. signed an informed consent form which was approved by the institutional review board of the respective medical center .

Exclusion Criteria:

1. Other invasive malignancies within 5 years except for adequately treated basal cell or squamous cell skin cancer, in situ carcinoma of the cervix;
2. Chemotherapy within 1 month;
3. Had received rituximab or other anti-CD20(+) monoclonal antibody treatment within 1 month before enrollment;
4. Had received rituximab or other anti-CD20(+) monoclonal antibody treatment 1 month ago but with ADA(+) before enrollment;
5. Blood concentration of Rituximab> 24 μg/ml prior to study entry;
6. Had received hematopoitic growth factor within 1 week prior to study entry;
7. Receipt of a live/attenuated vaccine within 4 weeks prior to the Screening Visit;
8. Recent major surgery (within 8 weeks prior to screening, excluding lymph node biopsy);
9. Peripheral or central nervous system disease;
10. Serious hematologic dysfunction (white blood cell count of <3.0×109/L; absolute neutrophil count of <1.5×109/L; platelet count of < 100×109/L; hemoglobin level of < 9.0 g/dL);
11. Hepatic dysfunction (total bilirubin level of > 1.5 × upper limit of normal (ULN); aspartate amino transferase (AST) and alanine amino transferase (ALT) levels of > 2.0 × ULN; alkaline phosphatase > 3.0 × ULN; renal dysfunction (serum creatinine level of > 1.5×ULN );
12. Abnormal thyroid function;
13. Seropositive for HIV , HCV antibody; seropositive for hepatitis B virus surface antigen (HBsAg). HBV DNA>1.0×103copies/ml;
14. Serious underlying medical conditions, could impair the ability of the patient to participate in the trial (including but not limited to ongoing active infection, uncontrolled diabetes mellitus, significant cardiac disease, uncontrolled angina, gastric ulcers, active autoimmune disease);
15. Pregnancy or breast feeding. For women of childbearing potential.
16. History of a severe allergic reaction or anaphylactic reaction to a biological agent or history of hypersensitivity to any component of the trial drug.
17. Subjects had a history of alcoholism or drug abuse;
18. Researchers think that do not fit into the group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) for HLX01 and rituximab concentrations | 91 days

SECONDARY OUTCOMES:
The Maximum Concentration (Cmax) of the HLX01 and rituximab | 91 days
Presence of Anti-Drug Antibodies against HLX01 | 91 days
Change from baseline of CD19+ B-cells | 91 days

REFERENCES:
- [Result] Shi Y, Zhang Q, Han X, Qin Y, Ke X, Su H, Liu L, Fu J, Jin J, Feng J, Hong X, Zhang X, Wu D, Jiang B, Dong X. Phase 1 studies comparing safety, tolerability, pharmacokinetics and pharmacodynamics of HLX01 (a rituximab biosimilar) to reference rituximab in Chinese patients with CD20-positive B-cell lymphoma. Chin J Cancer Res. 2021 Jun 30;33(3):405-416. doi: 10.21147/j.issn.1000-9604.2021.03.11. PMID 34321836